CLINICAL TRIAL: NCT07130734
Title: Digitally-Delivered Intervention to Prompt Physical Activity
Brief Title: Digital Intervention for Physical Activity
Acronym: DPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Christopher Brush, Assistant Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00000675
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Depression - Major Depressive Disorder; Anxiety; Stress
Keywords: Physical Activity; Digital Intervention; Depression; Mobile Application
MeSH Terms: conditions — Anxiety Disorders; Motor Activity; Depression

STUDY DESIGN:
Intervention Model Description: Between-subjects randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcomes assessor will be unaware of group assignment; research staff working for the investigator will perform randomization. Participants will know whether they are assigned to the digital physical activity or passive control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Intervention Group (Experimental): Participants allocated to this group will be instructed to download a Pathverse mobile application on their Apple or Android smartphone device. The Pathverse mobile application will be used to send participants daily push notifications to engage in physical activity of their choice. During on-boarding at pre-intervention, each participant will choose approximately five types of physical activity they find enjoyable that they would like to engage in throughout the four-week intervention. They will report on the physical activity they completed, along with the duration and intensity of each activity. Participants will have the choice of when they would like to receive their daily notifications on their smartphone device.
  Interventions: Behavioral: Digital Physical Activity
- Passive Control Group (No Intervention): Participants will be informed that their mental health will be monitored over four weeks as a control condition. After the study, they will be offered the digital PA intervention, if desired.

INTERVENTIONS:
Behavioral: Digital Physical Activity — The Pathverse mobile application platform will be downloaded on each participant's smartphone. Participants will be guided on how to download and use the application, as well as how to interact with the application during the intervention period. Participants will choose approximately five types of physical activity they enjoy before the intervention and will be prompted to complete these physical activities throughout the intervention. Participants will also self-report the duration and type of physical activity performed each day of the intervention.
  Arms: Digital Intervention Group

SUMMARY:
The present study will assess the effects of a four-week digitally delivered intervention on physical activity and depressive symptoms among adults experiencing at least moderate depressive symptoms. The main questions this research aims to answer are:

* Does a digitally-delivered intervention increase physical activity levels?
* Does a digitally-delivered intervention reduce symptoms of depression?

Researchers will compare an intervention promoting physical activity to a passive control (does not receive the intervention) group to see if the intervention reduces depressive symptoms and increases physical activity levels.

Participants will:

* Visit the laboratory at two separate time points before group assignment, separated by one week of physical activity monitoring
* Be randomly assigned to complete four weeks of a digital intervention prompting engagement in physical activity or have their mental health symptoms monitored over four weeks (i.e., passive control group)
* Visit the laboratory at two separate time points after the intervention, separated by one week of physical activity monitoring

DETAILED DESCRIPTION:
Procedures include four laboratory visits: two visits before the intervention and two visits after the intervention.

Participants will be randomly assigned to either four weeks of a digital intervention that prompts participants to engage in physical activity or a waitlist (passive) control condition. Participants will be randomized using a stratified approach using depressive symptoms and physical activity measured at pre-intervention as strata.

The digital intervention group will be instructed to download a Pathverse mobile application on their Apple or Android smartphone device. The Pathverse mobile application will be used as a research delivery platform that can send participants daily push notifications to engage in physical activity of their choice. During the second pre-intervention visit, each participant will select approximately five types of physical activity they find enjoyable that they would like to engage in over the four-week intervention. Participants will report on the physical activity they completed, along with the duration and intensity of each activity. Participants will have the choice of time of day as to when they would like to receive daily notifications on their device.

Members of the passive control group will be informed that their mental health will be monitored over four weeks as a control condition. After the study, they will be offered the digital PA intervention, if desired.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 19 and 40 years
* Verbally fluent in English (i.e., must be able to speak or understand English)
* No uncorrected visual or hearing impairment
* Moderate depressive symptoms or greater of at least 10 or higher on the Patient Health Questionnaire-8 screening instrument
* Eligible to participate in physical activity
* Physically inactive (i.e., engaging in less than 150 min of weekly moderate-to-vigorous physical activity)
* Owns an Apple or Android mobile device, willing to download the Pathverse app , and willing to keep the device on during the study period
* Not currently pregnant

Exclusion Criteria:

- Participants will not qualify for the current study if they do not meet the above inclusion criteria.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptoms | pre-intervention, at the two-week time point during the intervention, and immediately after the intervention
  Depression, Anxiety, and Stress Scale (DASS-21) will be used to assess changes in symptoms of depression. The DASS-21 includes 7 items that assess for depression. Total scores for depression range from 0-42, with higher scores indicating greater depression severity.
Moderate-to-vigorous physical activity | pre-intervention and immediately after the intervention
  Physical activity will be assessed using a wrist-worn accelerometer before and after the intervention. Physical activity outcomes will be calculated as amount of time spent in a specific intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- Kinesiology Building, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-09-12): https://cdn.clinicaltrials.gov/large-docs/34/NCT07130734/ICF_000.pdf